CLINICAL TRIAL: NCT06735196
Title: Profiling the Variation of Microbiome Along the Intestinal Tract Based on Sampling Capsule Endoscopy: a Feasibility and Safety Study
Brief Title: Profiling the Variation of Microbiome Along the Intestinal Tract Based on Sampling Capsule Endoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Clinical Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SCE-I
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers Only
Keywords: sampling capsule endoscopy; gut microorganisms; intestinal fluids; stool; saliva
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy volunteers (Other): After standard gastrointestinal preparation, healthy volunteers swallowed SCEs to collect intestinal fluids in different intestinal areas.
  Interventions: Device: sampling capsule endoscopy

INTERVENTIONS:
Device: sampling capsule endoscopy — Healthy volunteers swallowed SCEs to collect intestinal fluids in different intestinal areas. When SCEs excreted, the fluids inside SCEs would be collected for microbiome and metabolome analysis.

SUMMARY:
Intestinal flora and metabolites are associated with multiple systemic diseases. Current approaches for acquiring information regarding microbiota/metabolites have limitations. We aimed to develop a precise sampling capsule endoscopy (SCE) for the convenient, non-invasive, and accurate acquisition of digestive bioinformation for disease diagnosis and evaluation. The SCE was used for sampling jejunum, ileum, and colon content in healthy volunteers. The GI liquid was then used for microbiome profiling and metabolomics profiling. In this study, we aimed to describe the characteristics and functions of key microflora in the whole intestinal microenvironment of healthy volunteers.

DETAILED DESCRIPTION:
Gut microorganisms involved in human food digestion, immune system regulation, and protection against pathogens are critical in maintaining health. Gut microorganism dysbiosis influences the course of gastrointestinal disease and cardiovascular, neurological, metabolic diseases, and other disorders. Therefore, a deeper understanding of gut microorganisms is indispensable in researching human disorders. However, current sampling methods, including fecal microbial examination, breath hydrogen testing, and invasive endoscopy acquisition, fail to obtain local gut microbiome samples under its chemical environment in natural and unperturbed states. A comfortable, non-invasive, and precise regional intestinal fluid collection device is needed.

Recently, novel ingestible devices have collected intestinal fluids from animals' and humans' jejunum, ileum, and colon. Significant differences between bacteria and metabolites in the intestines versus stool have been identified, showing the spatiotemporal structure of the gastrointestinal microbiome and metabolome. Compared with saliva and stool samples, ingestible devices acquired samples in an environment resembling nature, which is more reliable in explaining the association between gut microorganisms dysbiosis and various disorders.

However, current ingestible sampling devices still have several limitations. Therefore, a novel sampling capsule endoscopy (SCE) system was developed. This novel SCE can precisely and efficiently acquire intestinal bio information through direct visualization under electric control. This study aims to collect fluids from different segments of the gastrointestinal tract using the SCE system to clarify the differences in the distribution of gut microorganisms in different areas in healthy volunteers and patients with inflammatory bowel disease or colon cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥18 years and ≤80 years;
2. American Society of Anesthesiologists (ASA) physical health risk level 1;
3. Good overall health, no clinically significant medical history;
4. No clinically significant signs were found in the physical examination;
5. For women of fertility, the urine pregnancy test was negative within 7 days after the screening visit, and they were willing to take contraceptive measures throughout the study;
6. Willing to provide blood samples, stool samples, urine samples, saliva samples, and intestinal fluid samples, and agree that the samples provided will be stored for a long time and used for research purposes.
7. Agree to avoid strenuous activities during the participation in this clinical trial;
8. Agree to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

1. Patients with digestive tract diseases such as cancer, inflammatory bowel disease, achalasia, esophageal diverticulum, etc.;
2. Patients who have participated in other clinical trials within three months or are currently participating in other clinical trials;
3. Patients currently use medication for other diseases or plan to use medication for treatment;
4. Patients who have used antibiotics within three months;
5. Patients with known or suspected gastrointestinal obstruction, stenosis, diverticulum, and fistula;
6. Patients with swallowing disorders;
7. Pregnant or lactating women or women who plan to become pregnant within 30 days of the visit period;
8. Patients who are not suitable for surgery or refuse to undergo any abdominal surgery (once the capsule is retained, it cannot be removed by surgery);
9. Patients with any form of active substance abuse or dependence (including drug or alcohol abuse), any unstable physical or mental illness, any malignant lesions in any location or system, or any chronic disease that the researcher believes may interfere with the study;
10. The researcher believes any other factors are unsuitable for selection or affect the subject's participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The feasibility of sampling capsule endoscopy system in collecting fluids from different intestinal segments in healthy volunteers | two weeks
  The total successful rate of SCE in sampling fluids in intestinal segments. A successful sampling procedure conducted by SCE was defined when the following conditions were met simultaneously: 1) accurately recognization of target intestinal areas. 2) the intestinal liquid can be successfully collected in the sampling chamber.

SECONDARY OUTCOMES:
Standard gastrointestinal preparation procedure | two week
  To select the best standard gastrointestinal preparation procedure which makes the visualization score under SCE graded as the best (on a scale of 1 to 5; 1, the worst; 5, the best) .
Sampling time | two weeks
  The total time for sampling intestinal fluids of a SCE.
Sampling volume | two weeks
  The overall volume of samples obtained by a SCE during a single examination.
Number of sampling times | two weeks
  Times we tried to sample during a single SCE examination.
Safety analysis | from enrollment to the end of follow-up at 30 days
  All adverse events occurring during the study

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Doctor, Principal Investigator — First Affiliated Hospital of Naval Medical University (Changhai Hospital)
Locations (1):
- First Affiliated Hospital of Naval Medical University (Changhai Hospital), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zoetendal EG, Raes J, van den Bogert B, Arumugam M, Booijink CC, Troost FJ, Bork P, Wels M, de Vos WM, Kleerebezem M. The human small intestinal microbiota is driven by rapid uptake and conversion of simple carbohydrates. ISME J. 2012 Jul;6(7):1415-26. doi: 10.1038/ismej.2011.212. Epub 2012 Jan 19. PMID 22258098
- [Background] Kastl AJ Jr, Terry NA, Wu GD, Albenberg LG. The Structure and Function of the Human Small Intestinal Microbiota: Current Understanding and Future Directions. Cell Mol Gastroenterol Hepatol. 2020;9(1):33-45. doi: 10.1016/j.jcmgh.2019.07.006. Epub 2019 Jul 22. PMID 31344510
- [Background] Ding Z, Wang W, Zhang K, Ming F, Yangdai T, Xu T, Shi H, Bao Y, Yao H, Peng H, Han C, Jiang W, Liu J, Hou X, Lin R. Novel scheme for non-invasive gut bioinformation acquisition with a magnetically controlled sampling capsule endoscope. Gut. 2021 Dec;70(12):2297-2306. doi: 10.1136/gutjnl-2020-322465. Epub 2021 Jan 15. PMID 33452177